CLINICAL TRIAL: NCT01514110
Title: Phase I/II Study of Paclitaxel / Carboplatin / RAD001 as First Line Therapy for Advanced Adenocarcinoma of the Stomach
Brief Title: Gastric Cancer RAD001 Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAT006
Record Dates: First submitted 2011-11-22; First posted 2012-01-20 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Everolimus; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — Pharmacology of RAD001 as a combination partner for conventional agents.
  Other Names: RAD001 with Paclitaxel 175 mg/m2 and carboplatin (AUC=5) on Day 1, every 3 weeks until PD

SUMMARY:
The purpose of this study is to determine dose limiting toxicities (DLT) and maximum tolerated dose (MTD) of RAD001, as well as to assess tumor response and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the stomach. Patients who have adenocarcinoma of the gastroesophageal junction will be eligible if the majority of the tumor bulk is below the junction.
* Metastatic or Loco-regionally advanced disease
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT /MRI scan. See section 11.2 for the evaluation of measurable disease.
* Age >= 18 years.
* Life expectancy of greater than 12 weeks.
* ECOG performance status <= 2 (Karnofsky >= 60%).

Exclusion Criteria:

* Patients who have received more than one line of palliative chemotherapy are allowed, provided that (i) the prior chemotherapy does not contain taxane, cisplatin or carboplatin; (ii) 4 weeks have elapsed prior to the start of the current study treatment, and that (iii) they have recovered from adverse events due to previous treatment [except alopecia].
* Patients who have had radiotherapy or major surgery within 4 weeks prior to entering the study or those who have not recovered from adverse events due to treatment administered more than 4 weeks earlier.
* Patients who are on CYP3A4 modifiers are excluded from the study
* Patients with known brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RAD001.

Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, congestive heart failure related to primary cardiac disease, a condition requiring anti-arrhythmic therapy, ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to the trial entry.

* Patients with severe concurrent medical illness such as severe impairment of lung function should be excluded from studies of RAD001.
* Uncontrolled intercurrent such as, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Poorly controlled diabetes mellitus
* High LDL cholesterol or triglyceride level
* Pre-existing neuropathy of >= grade 2
* Patients with a history of second malignancies are eligible they have been disease free for at least 5 years and are deemed by the investigator to be at low risk of recurrence. Par8entswith the following cancers are eligible if diagnosed and treated within the past 5 years: cervical carcinoma in situ, melanoma in situ, and basal cell or squamous cell carcinoma of the skin
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01-23 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
to determine the Maximum tolerated dose and dose limiting toxicity of RAD001 in combination with paclitaxel and carboplatin | 2 years

SECONDARY OUTCOMES:
Toxicity of combination Paclitaxel/carboplatin/RAD001 in advanced adenocarcinoma of the stomach and gastroesophageal junction | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Yeo, MD, FRCP, Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong